CLINICAL TRIAL: NCT07181343
Title: A Study to Evaluate the Pharmacokinetics of Drospirenone and Ethinyl Estradiol Tablets (Yasmin®) When Co-administered With HS-10374 Tablets
Brief Title: A Drug-Drug Interaction Study Between HS-10374 Tablets and Drospirenone and Ethinyl Estradiol Tablets(Yasmin®)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hansoh BioMedical R&D Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HS-10374-118
Record Dates: First submitted 2025-08-20; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Psoriasis (PsO)
MeSH Terms: conditions — Psoriasis | interventions — drospirenone; Ethinyl Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HS-10374 + Drospirenone and Ethinyl Estradiol (Experimental)
  Interventions: Drug: HS-10374 tablets; Drug: Drospirenone and Ethinyl Estradiol tablets

INTERVENTIONS:
Drug: HS-10374 tablets — From Day 8 to Day 19, participants will orally take HS-10374 Tablets 12 mg（6 mg×2） once daily under fasting conditions
Drug: Drospirenone and Ethinyl Estradiol tablets — On Day 1 and Day 14, participants will orally take one tablet of Drospirenone and Ethinylestradiol Tablets under fasting conditions.

SUMMARY:
This trial is a single-center, open-label, fixed-sequence, self-controlled clinical study to evaluate Drug-Drug Interaction Between HS-10374 Tablets and Drospirenone and Ethinyl Estradiol Tablets (Yasmin®)

DETAILED DESCRIPTION:
This trial is a single-center, open-label, fixed-sequence, self-controlled clinical study. On Day 1 and Day 14, participants will orally take one tablet of Drospirenone and Ethinylestradiol Tablets (containing Drospirenone 3 mg and Ethinylestradiol 0.03 mg) under fasting conditions. From Day 8 to Day 19, participants will orally take HS-10374 Tablets 12 mg once daily under fasting conditions. Both drugs should be administered with approximately 240 mL of water.

ELIGIBILITY:
Inclusion Criteria:

* Participants who sign the informed consent form before the trial, fully understand the trial content, procedures, and potential adverse reactions, and voluntarily commit to complying with all trial requirements.
* Healthy female participants aged 18 to 40 years (inclusive), with age calculated based on the date of signing the informed consent.
* Participants weighing ≥45 kg, with a body mass index (BMI) ranging from 19.0 to 26.0 kg/m² (inclusive). BMI = weight (kg) / height² (m²).
* Participants who agree to abstain from conception/donation of oocytes and practice complete abstinence from signing the informed consent until 40 days after the last dose.

Exclusion Criteria:

* Participants with clinically significant abnormalities in physical examination, vital signs, ECG, clinical laboratory tests, abdominal ultrasound, gynecological color ultrasound, or breast color Doppler ultrasound, as judged by the investigator.
* Positive results for any of the following during screening: Hepatitis B surface antigen (HBsAg), hepatitis C antibody, HIV antibody/p24 antigen, or Treponema pallidum antibody.
* Screening values exceeding 1.5×ULN for ALT, AST, or creatine kinase (CK), with clinical significance per investigator assessment.
* Screening serum creatinine >1×ULN, judged clinically significant by the investigator.
* QT interval prolongation on 12-lead ECG during screening (QTcF ≥470 ms).
* History of myopathy or rhabdomyolysis.
* Severe pre-existing or current diseases affecting the nervous, psychiatric, digestive, circulatory, respiratory, urinary, cardiovascular, or immune systems-or any newly diagnosed condition prior to dosing-deemed by the investigator to contraindicate participation; including history of gastrointestinal disorders (e.g., gastric ulcer, reflux esophagitis).
* History of tuberculosis (TB).
* Current or previous history of: Venous thromboembolism (e.g., deep vein thrombosis, pulmonary embolism), Cerebrovascular disorders, Coronary artery disease, hypertension, Thrombogenic cardiac valvulopathy or rhythm disorders (e.g., subacute bacterial endocarditis with valvular disease, atrial fibrillation), Hereditary/acquired hypercoagulable states (e.g., Factor V Leiden mutation family history), Diabetes with vascular complications, Headaches with focal neurological symptoms, Migraine (with or without aura), Cholestatic jaundice and/or pruritus during prior hormone therapy.
* Current or previous renal impairment or adrenal insufficiency.
* Undiagnosed abnormal uterine/vaginal bleeding.
* Current or previous estrogen/progestin-sensitive cancers (e.g., breast cancer).
* Benign/malignant liver tumors or severe liver disease with safety risks per investigator judgment.
* Active/latent TB infection during screening, assessed by: T-SPOT.TB (interferon-gamma release assay),Chest X-ray. Exclusion if: Chest X-ray shows TB lesions OR T-SPOT.TB positive.
* Severe infections ≤30 days before screening (e.g., cellulitis, pneumonia, sepsis) OR herpes zoster within 3 months prior.
* Participants who have undergone surgery affecting drug absorption, distribution, metabolism, or excretion, deemed ineligible by the investigator.
* Individuals with a history of hypersensitivity or allergic predisposition (e.g., to pollen, ≥2 drugs/foods), or known allergy to: Active ingredients/excipients of the investigational products (Drospirenone and Ethinylestradiol Tablets & HS-10374 Tablets), Other Janus Kinase (JAK) inhibitors.
* Participation in any other clinical trial involving investigational drugs/devices within 3 months prior to screening .
* Blood donation or significant blood loss (>400 mL) within 3 months before screening, or plans to donate blood during the trial or within 1 month after completion .
* Ingestion of grapefruit or grapefruit products within 48 hours before the first dose of investigational products .
* Excessive consumption of tea, coffee, or caffeine-containing beverages (>8 cups/day on average; 1 cup=200 mL) within 3 months prior to screening .
* Participants who smoked ≥1 cigarette/day within 3 months before screening, were unable to quit tobacco products during the trial, or tested positive for nicotine.
* Participants who drank alcohol frequently (>14 units/week, 1 unit =14 g alcohol) within 3 months before screening, couldn't stop using alcohol during the trial, or tested positive for alcohol in breath tests.
* Participants who used alcohol-containing products within 24 h before taking the test drug or had a positive alcohol breath test result.
* Participants with a history of drug abuse, dependence, or illicit drug use within 5 years before screening, or tested positive for drug abuse in urine tests.
* Participants who used drugs affecting liver metabolic enzymes (CYP3A, CYP1A2, CYP2D6, CYP2B6) or P-gp/BCRP activity, HIV/HCV protease inhibitors, non-nucleoside reverse transcriptase inhibitors, or hormonal drugs within 30 days before the first test drug dose.
* Participants who used long-acting estrogen/progestin injectables or implants within 12 months before the first dose, or transdermal contraceptives or intrauterine devices with hormones within 3 months before enrollment.
* Participants who used drugs altering gastric pH (e.g., rebamipide, omeprazole, lansoprazole, ranitidine, aluminum hydroxide) within 30 days before screening.
* Participants who used prescription drugs, OTC drugs, herbs, or health products (excluding local-acting topical agents) within 14 days before screening.
* Participants who used vaccines within 14 days before screening or planned to use them during or within two weeks after the trial.
* Participants who tested positive for pregnancy or were breastfeeding at screening.
* Participants who had unprotected sex within 14 days before screening.
* Participants unable to tolerate venipuncture/indwelling needle blood collection or with a history of fainting at the sight of blood.
* Participants unlikely to complete the trial for other reasons or deemed unsuitable by the investigator.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2025-05-28 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-08-19 (Actual)

PRIMARY OUTCOMES:
Evaluation of PK parameters of drospirenone and ethinylestradiol when used alone or in combination with HS-10374: Cmax | up to Day 20
  Maximum concentration
Evaluation of PK parameters of drospirenone and ethinylestradiol when used alone or in combination with HS-10374: AUC0-t | up to Day 20
  Area under the plasma concentration-time curve fom time 0 to last time of quantifiable concentration
Evaluation of PK parameters of drospirenone and ethinylestradiol when used alone or in combination with HS-10374: AUC0-24 h | up to Day 20
  Area under the plasma concentration-time curve fom time 0 to 24 h of quantifiable concentration
Evaluation of PK parameters of drospirenone and ethinylestradiol when used alone or in combination with HS-10374: AUC0-∞ | up to Day 20
  Area under the plasma concentration-time curve from time 0 extrapolated to infinite time

SECONDARY OUTCOMES:
Evaluation of PK parameters of drospirenone and ethinylestradiol when used alone or in combination with HS-10374: Tmax | up to Day 20
  Time to maximum concentration.
Evaluation of PK parameters of drospirenone and ethinylestradiol when used alone or in combination with HS-10374: t1/2z | up to Day 20
  Elimination half-life
Evaluation of PK parameters of drospirenone and ethinylestradiol when used alone or in combination with HS-10374: λz | up to Day 20
  Elimination rate constant.
Evaluation of PK parameters of drospirenone and ethinylestradiol when used alone or in combination with HS-10374: CLz/F | up to Day 20
  Plasma clearance.
Evaluation of PK parameters of drospirenone and ethinylestradiol when used alone or in combination with HS-10374: Vz/F | up to Day 20
  Apparent volume of distribution
Evaluation of PK parameters of drospirenone and ethinylestradiol when used alone or in combination with HS-10374: MRT0-t | up to Day 20
  Mean Residence Time from 0-t
Evaluation of PK parameters of drospirenone and ethinylestradiol when used alone or in combination with HS-10374: MRT0-∞ | up to Day 20
  Mean Residence Time from 0-∞
Evaluation of the pharmacokinetic characteristics of HS-10374 after multiple dosing：Cmax | up to Day 20
  Maximum concentration
Evaluation of the pharmacokinetic characteristics of HS-10374 after multiple dosing: Cmin | up to Day 20
  Minimum concentration
Evaluation of the pharmacokinetic characteristics of HS-10374 after multiple dosing: Cav | up to Day 20
  Steady State Concentration
Evaluation of the pharmacokinetic characteristics of HS-10374 after multiple dosing: AUC0-24h | up to Day 20
  Area under the plasma concentration-time curve fom time 0 to 24 h of quantifiable concentration
Evaluation of the pharmacokinetic characteristics of HS-10374 after multiple dosing: Tmax | up to Day 20
  Time to maximum concentration
Evaluation of the pharmacokinetic characteristics of HS-10374 after multiple dosing: t1/2z | up to Day 20
  Elimination half-life
Evaluation of the safety after single oral administration of HS-10374 tablets and drospirenone/ethinylestradiol tablets in healthy participants | through study completion, an average of 1 month
  Frequency of Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China